CLINICAL TRIAL: NCT07017452
Title: Methoxyflurane + Lorazepam + Percocet (Per os) vs Deep Intravenous Sedation: A Non-inferiority Randomized Controlled Trial to Assess the Efficacy and Safety During Convective Radiofrequency Water Vapor Thermal Therapy (REZUM) for Benign Prostate Hyperplasia
Brief Title: Trial to Assess the Efficacy and Safety During Convective Radiofrequency Water Vapor Thermal Therapy (REZUM) for Benign Prostate Hyperplasia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Premal Patel, MD, Assistant Professor, Department of Surgery. Director, Undergraduate Urologic Medical Education, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS27031
Record Dates: First submitted 2025-05-01; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Benign Prostate Hypertrophy(BPH)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — oxycodone-acetaminophen; Lorazepam; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: Single-centered, unblinded, randomized controlled trial. Two arms, one is the intervention arm which will receive Penthrox with a combination of Percocet and Lorazepam. The control arm will receive the standard of care during the rezum procedure which is deep IV sedation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention arm-Penthrox (Experimental): Participants can begin using penthrox 10 minutes prior to procedure start, given its median onset time of 5 minutes
  Interventions: Drug: Methoxyflurane - Penthrox; Drug: Percocet Pill; Drug: Lorazepam (drug)
- Control arm (Placebo Comparator): Patients will receive standard of care during their rezum procedure which consists of deep IV sedation.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Methoxyflurane - Penthrox — Penthrox is a brand name for a drug called methoxyflurane. It is an inhaled analgesic (pain-relieving) agent used primarily for the relief of moderate to severe pain, typically in emergency medical situations or during minor medical procedures. Penthrox is administered by inhaling the vapors through a hand-held inhaler device. It acts quickly to provide pain relief and has a relatively short duration of action.
  Arms: Intervention arm-Penthrox
Other: Control — This intervention will be the control group only, receiving deep IV sedation.
  Arms: Control arm
Drug: Percocet Pill — Percocet will be given in conjunction with methoxyfluorane and lorazepam
  Arms: Intervention arm-Penthrox
Drug: Lorazepam (drug) — Lorazepam will be given in conjunction with penthrox and percocet.
  Arms: Intervention arm-Penthrox

SUMMARY:
The primary aim of the study is to show that methoxyflurane-lorazepam-percocet combination administrated 'per os' is non inferior to deep intravenous sedation in achieving analgesia during Rezum convective radiofrequency water vapor thermal therapy for the management of benign prostate hyperplasia (BPH). We propose to conduct a single-centered, unblinded, randomized controlled trial designed after consulting ICH Guidelines for Good Clinical Practice as well the regulations set by the Biomedical Research Ethics Board, University of Manitoba.

DETAILED DESCRIPTION:
Participants who belong to the experimental arm will be given a single 'per os' dose of percocet (325mg acetaminophen + 7.5mg oxycodone) and lorazepam 1 mg, 30 minutes prior to the procedure. Patients will receive education on how to use the Penthrox inhaler device. Inside the operating room, the subject would self-inhale the methoxyflurane 5 minutes prior to the procedure. All these steps will be supervised by the clinical research nurse. Each participant will be administered with 3ml of methoxyflurane which is poured into the inhaler. Participants who were randomized to the control arm will receive deep intravenous sedation under the supervision of a trained anesthetist. A combination of midazolam, ketamine, remifentanil and propofol will be administered using an intravenous line. The quantity of these medications will be calculated by the anesthetist based on clinical judgement and also takes into account the physical characteristic of the subject. Both the groups receive the same Rezum water vapor therapy and the number of Rezum injections depends on the clinical judgement of the urologist performing the procedure. Immediately, post the procedure, the self-reported pain of the patient will be recoded using the NRS. A phone call follow-up would be done the following day to record any adverse events caused due to the procedure. Four weeks post the procedure, a phone call follow-up would be done to understand the patient satisfaction after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide an informed consent.
* Age ≥ 18 years
* Biological males identified with male sexual organs.
* Scheduled for convective radiofrequency water vapor thermal therapy (REZUM) for the management of benign prostate hyperplasia.

Exclusion Criteria:

* Concomitant use of nephrotoxic and/or hepatoxic agents.
* Use of ≥ 6 ml Penthrox withing the previous 3 weeks.
* Known allergies and/or adverse events due to penthrox, other halogenated anesthetics, percocet (oxycodone + acetaminophen), lorazepam, lidocaine, midazolam, ketamine, remifentanil and propofol
* History of genetic susceptibility to malignant hyperthermia.
* Presence of clinically significant respiratory depression, cardiovascular instability, renal or hepatic impairment
* Altered level of consciousness due to any cause.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Post-Procedural Pain | Immediately post-procedure
  Post procedural pain measured using the Numeric Rating Scale for pain. Higher scores on this measurement indicate worser outcomes. Maximum value of 10 and a minimum value of 10 can be reported on this scale.

SECONDARY OUTCOMES:
Safety of Procedure | At time of procedure and post-procedure
  The safety of combination vs deep intravenous sedation during Rezum will be measured by accounting for adverse event encountered during the procedure.
Cost-effectiveness, | 1 month post-procedure
  We will compare the costs associated with the procedure in both arms to see if there is any difference.
Anxiety levels | Pre-Procedure on day of procedure
  We will measure anxiety levels using the Amsterdam Pre-Operative Anxiety and Information Scale (APAIS). Higher scores indicate worser outcomes. Maximum value of 30 and a minimum value of 0. It is a 6 part questionnaire which each question is given on a likert scale from 1-5
Patient satisfaction | Immediately post-procedure
  We will measure patient satisfaction using a likert scale single question patient satisfaction questionnaire. (higher scores indicate better outcomes). Maximum value of 5 and a minimum value of 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Men's Health Clinic Manitoba, Winnipeg, Manitoba, Canada